CLINICAL TRIAL: NCT07129811
Title: The Effect of Ultrasound-Guided Stellate Ganglion Block on Pain, Functionality, and Quality of Life in Type 1 Complex Regional Pain Syndrome in Stroke Patients
Brief Title: Stellate Ganglion Block in Complex Regional Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Seher KALIÇ, Principle Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TABED 1-24-804; Ankara Bilkent City Hospital (Other: Ankara Bilkent City Hospital)
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Stellate Ganglion Block
Keywords: Stroke; chronic pain; Complex regional pain syndrome
MeSH Terms: conditions — Stroke; Chronic Pain; Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher conducting the evaluations will not know the group the patient will be assigned to. The other researcher will determine which group the patient will be assigned to through randomization and will perform the intervention if the patient is in the stellate ganglion group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellat Group (Active Comparator): In group 1, stellate ganglion blockade will be applied in addition to conventional physical therapy.
  Interventions: Procedure: Stellate Ganglion Block
- Only Physical Therapy Group (No Intervention): Group 2 will receive only conventional physical therapy and exercise therapy

INTERVENTIONS:
Procedure: Stellate Ganglion Block — The stellate ganglion is located in front of the anterior tubercle of the C6 vertebra. An ultrasound-guided intervention will be performed from the affected side and 2 cc of 1% lidocaine will be injected.
  Arms: Stellat Group

SUMMARY:
The aim was to investigate the effect of Stellate Ganglion Blockade, which will be applied in addition to conventional physical therapy, on pain and functionality in patients with poststroke complex regional pain syndrome.

DETAILED DESCRIPTION:
Post-stroke complex regional pain syndrome (CRPS) is relatively common in hemiplegic upper extremity. Complex regional Pain Syndrome Type 1 is often seen without any nerve damage especially post-stroke. This musculoskeletal disorder usually effects motor improvement, quality of life and Daily living activities. Besides Presence of CRPS is thought to be challenging on the way of rehabilitation process. However, disproportionate sympthatic nervous system activation, disinhibition of the descenden neuronal pathways are the mechanisms thought to be taken place in the etiopathogenesis of CRPS, it still remains unclear. Pharmacological agents, Physical Therapy techniques, exercise and injections are used to treat CRPS. Therefore post-stroke patients have co-morbidities and multi-drug usage, it should be take into account to treat them with physical therapy agents and interventional procedures. Stellat ganglion blockade is an interventional technique that is used to break the vicious circle of symphatetic activation of upper extremity in CRPS. However to the best of our knowledge there are not any study that evaluates the effect of stellat ganglion Blockade on CPRS combining conventional physical therapy. Total of 32 patients with post-stroke CPRS are going to be participated in the study. Patients are going to be divided into two groups. Group 1 is going to receive both onventional physical therapy, exercise (10 sessions) and stellat ganglion blockade and Group 2 is going to receive just conventional physical therapy program and exercise therapy (10 sessions). Participants are going to evaluate before treatment, 2 weeks and 12 weeks after the end of the therapy sessions. Visual analog scale (VAS), Brunnstroom stages of stroke recovery (BSSR), Fugl-meyer (FMUE) and Stroke spesific quality of life (SSQoL) are used to evaluate pain, functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer male and female patients aged 18-75
* Diagnosed with Complex Regional Pain Syndrome according to the IASP 2012 Diagnostic Criteria
* Patient's pain level must be VAS >4

Exclusion Criteria:

* Presence of existing neurological diseases other than rheumatic diseases and stroke
* General impairment
* Conditions that would constitute a contraindication to application, such as an open wound or sensory deficit in the application area
* Presence of active infection
* Presence of malignancy
* Cognitive dysfunction (mini mental test result <23)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before treatment, 2 weeks and 12 weeks after the end of sessions
  Ten-cm VAS was used as a self-report measure for lower back pain intensity. Self reported pain measurement score is between 0-10 and higher scores indicates higher pain severity.

SECONDARY OUTCOMES:
Brunnstroom stages of stroke recovery (BSSR) | before treatment, 2 weeks and 12 weeks after the end of the therapy sessions
  The BSSR is used to evaluate the motor development of the hemiplegic upper extremity, lower extremity and hand in stroke patients using a staging system from 1 (flask) to 6 (normal motor function).
Fugl-Meyer Upper Extremity (FMUE) Scale | before treatment, 2 weeks and 12 weeks after the end of the therapy sessions
  The FMUE scale is a stroke- specific, performance-based measure of sensory motor impairment consisting of 33 items, each scored on a scale of 0 to 2. Higher scores signify a lower level of impairment.
Stroke Specific Quality of Life scale (SS-QOL). | before treatment, 2 weeks and 12 weeks after the end of the therapy sessions
  The SS-QOL is a questionnaire used to evaluate independence in ADL in patients with stroke, social role within the family and community and quality of life (QOL). It consists of 49 questions scored between one and five giving a total score between 49 and 245. Higher scores indicate better QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Its going to be shared after the end of study

REFERENCES:
- [Background] Yoo SD, Jung SS, Kim HS, Yun DH, Kim DH, Chon J, Hong DW. Efficacy of ultrasonography guided stellate ganglion blockade in the stroke patients with complex regional pain syndrome. Ann Rehabil Med. 2012 Oct;36(5):633-9. doi: 10.5535/arm.2012.36.5.633. Epub 2012 Oct 31. PMID 23185727
- [Background] Narouze S. Ultrasound-guided stellate ganglion block: safety and efficacy. Curr Pain Headache Rep. 2014 Jun;18(6):424. doi: 10.1007/s11916-014-0424-5. PMID 24760493
- [Background] Harden RN, McCabe CS, Goebel A, Massey M, Suvar T, Grieve S, Bruehl S. Complex Regional Pain Syndrome: Practical Diagnostic and Treatment Guidelines, 5th Edition. Pain Med. 2022 Jun 10;23(Suppl 1):S1-S53. doi: 10.1093/pm/pnac046. PMID 35687369
- [Background] Altas EU, Onat SS, Konak HE, Polat CS. Post-stroke complex regional pain syndrome and related factors: Experiences from a tertiary rehabilitation center. J Stroke Cerebrovasc Dis. 2020 Sep;29(9):104995. doi: 10.1016/j.jstrokecerebrovasdis.2020.104995. Epub 2020 Jul 3. PMID 32807418